CLINICAL TRIAL: NCT04035941
Title: The Cycle Nation Project: A Workplace Intervention to Increase the Number of People Cycling Regularly (Phase 2: Feasibility)
Brief Title: The Cycle Nation Project (Phase 2: Feasibility)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Glasgow (Other)
Collaborators: University of Edinburgh (Other)
Responsible Party: Principal Investigator, Professor Jason Gill, Professor of Cardiometabolic Health, University of Glasgow
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 200180138
Record Dates: First submitted 2019-07-19; First posted 2019-07-29 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Health Behavior
Keywords: physical activity; cycling
MeSH Terms: conditions — Health Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: Study design: A before-and-after feasibility study with follow up to six months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Feasibility (Experimental): The cycle training intervention group
  Interventions: Behavioral: Cycle Nation Multicomponent Intervention

INTERVENTIONS:
Behavioral: Cycle Nation Multicomponent Intervention — This intervention group will receive 4 elements:
  1. Practical skills programme: a workplace-based programme covering basic cycling skills, delivered by trained 'cycle champions' - HSBC staff members.
  2. Cycle provision scheme: participants will have the opportunity to have their own bicycles serviced or obtain a loaned bike or e-bike from local bike shops before the start of the programme.
  3. Cycle-friendly workplace culture: all offices taking part will have a minimum of secure bike parking facilities as part of an ongoing roll-out of cycle infrastructure across HSBC UK offices.
  4. Our Cycle Hub app: an adapted version of an existing HSBC app including route planning, goal setting and practical skills videos, as well as supportive social interaction among participants.

SUMMARY:
Interventions to increase the number of people cycling regularly are likely to induce a range of health and societal benefits, including reduced incidence of heart disease, cancer and obesity, improved mental health and well-being, and reduced road congestion and air pollution. They are also likely to provide tangible financial and in-kind benefits to employers and society, through reduced workforce absenteeism, increased productivity and decreased use of NHS resources. However, increasing the number of people cycling regularly is complex and interventions undertaken to date have only been modestly successful. Thus, to induce a step-change in the number of people cycling in the United Kingdom (UK), in line with British Cycling and HSBC UK's stated aim of getting two million more people on bikes, new approaches are needed.

The research team have been working with staff and management at British Cycling and HSBC to co-develop a novel, multi-component intervention for delivery at HSBC offices to increase the number of employees cycling regularly. The intervention has four main components: 1) a six (intermediate) or nine (foundation) week practical skills programme; 2) cycle provision (tune-up/loan/subsidised purchase) schemes; 3) establishment of a cycle-friendly workplace culture; 4) a cycle app. The purpose of this study is to test the feasibility of this intervention in a before-and-after study in four HSBC offices around the UK.

DETAILED DESCRIPTION:
Objective: To assess the feasibility of the novel multicomponent workplace cycling intervention that aims to support more employees to cycle regularly. There are eight related research questions:

1. Can sufficient (~20-30) employees per HSBC office be recruited to take part in the intervention?
2. Can participants be retained in the study for up to three months?
3. To what extent do participants receive the intervention as intended (exposure)?
4. To what extent is the intervention acceptable to participants, those leading the intervention (local cycle champions), local HSBC office management and local bike providers?
5. How feasible and acceptable is it to conduct a suite of measurements, including self-report questionnaires, objective physical activity and blood biomarkers of cardiovascular disease, in this setting?
6. Does the intervention have potential to increase cycling and cycle journeys (likely primary outcomes in a future RCT)?
7. To what extent do participants improve on a range of behavioural, psychological, clinical and work-related outcomes?
8. Does the intervention have potential to be cost-effective, and what are the range of cost and benefit outcomes that are to be considered?

Setting and Participants: The study will be conducted at four HSBC offices across the UK, which have some degree of on-site cycle infrastructure (e.g. secure bike racks, showers, lockers). At each office, up to 40 participants will be recruited to either the foundation (nine-week) or intermediate (six-week) practical skills programme (up to 160 participants in total across the four sites). Participants will be self-identified infrequent cyclists (currently cycle less than once per month or not at all) aged 18 years or over who are current HSBC employees.

Interventions:

The intervention has four main components.

1. Practical skills programme: this has two versions - a core six-week programme (intermediate), with an additional three weeks (nine weeks in total - foundation) covering basic cycling skills. It is designed to be delivered at HSBC offices by trained 'cycle champions' - ideally HSBC staff members. Each session includes group-based learning activities and in-saddle, off- and on-road practical cycle training. Participants will receive information delivered simply in handbook format with a "toolkit" of skills and behaviour change techniques (e.g. goal setting) participants can apply to increase their cycling and maintain this long-term.
2. Cycle provision scheme: participants will have the opportunity to have their own bicycles serviced or obtain a loaned bike or e-bike from local bike shops before the start of the programme. At the end of the programme, participants will be given support and advice to take part in the HSBC subsidised cycle purchase bike to work scheme.
3. Cycle-friendly workplace culture: all of the HSBC offices taking part in the study will have a minimum of secure bike locks as part of an ongoing roll-out of cycle infrastructure across HSBC UK offices. During training, the cycle champion will be asked to identify (and subsequently implement) other cycle-friendly features (e.g. availability of cycle tools and spares, flexible hours to avoid peak commuter traffic, flexible dress code, altruistic reward scheme for cycling).
4. Our Cycle Hub app: an adapted version of an existing HSBC app including route planning, goal setting and practical skills videos, as well as supportive social interaction among participants.

Outcomes:

The feasibility study will assess: recruitment, retention, adherence, feasibility of delivery of all components, fidelity to intervention protocol, acceptability (to participants and cycle champions, other staff in the office who are not doing the practical skills programme but are exposed to the cycle-friendly culture, HSBC office managers and bike providers), and likely primary outcomes of any future randomised controlled trial (RCT) - number of people cycling regularly (both monthly and weekly) and number of cycling journeys for transport or leisure in the last month, both self-reported. The investigators will also assess likely secondary outcomes in a future RCT at baseline, 9 weeks, and 13 weeks.

1. behavioural - objectively-measured cycling and other physical activity (using the activPAL device and a new algorithm specifically-developed to detect cycling) and self-reported cycling activity, modes of transport, physical activity, sedentary behaviour, sleep, dietary intake.
2. psychological - self-reported motivation, autonomy, competence, relatedness and perceptions of safety in relation to cycling, wellbeing, self-esteem, vitality, quality of life and perceived general physical health.
3. work-related - productivity, job satisfaction, occupational stress, absenteeism and presenteeism.
4. clinical - objectively-measured weight, height, BMI, waist circumference, diastolic and systolic blood pressure. Cardio-metabolic disease risk biomarkers related to glucose, insulin, HbA1c, lipids and liver function will be assessed at baseline and 13 weeks only (opt in).

Participant characteristics (e.g. date of birth, gender, postcode of residence, marital status, education, smoking status, alcohol consumption, job description) will be recorded at baseline only. Extent of delivery, acceptability and perceived utility of programme components (practical skills programme components, bike provision, cycle-friendly culture and cycle app), and acceptability of the study procedures will be assessed at follow up only. Adverse events and injury will be assessed at all time points. Health economists will work with HSBC head office staff to identify available sources of cost and benefit data throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Any staff members who currently cycle less than once per month or not at all

Exclusion Criteria:

* Staff members who currently cycle more than once per month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-08-05 (Estimated); Primary Completion 2020-04-30 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of intervention delivery: Investigator conducted session observations | 9 weeks
  To measure the feasibility of delivery of all cycle training components by investigator conducted session observations.
Feasibility of intervention delivery: Investigator conducted interviews | 9 weeks
  To measure the feasibility of delivery of all cycle training components by investigator conducted interviews with cycle champions.
Cycling behaviour | Change from baseline to 13 weeks
  Self reported number of people cycling regularly (both monthly and weekly) and number of cycling journeys for transport or leisure in the last month.
Participant and Cycle Champion recruitment | Conducted pre baseline
  Measeurement of the recruitment of participants and cycle champions.
Participant and Cycle Champion retention | Change from baseline to 9 weeks
  Measurement of the number of participants and cycle champions who undertake the training course to completion, as well as participant drop-out
Participant adherence to the cycle training course | Through study completion to 9 weeks
  Measurement of participant attendance to training sessions
Cycle Champion interviews: acceptability of cycle training course delivery | 9 weeks
  Interview measured acceptability of all elements of intervention delivery (cycle champions)
Participant questionnaire: Likert scale of training course acceptability | 9 weeks
  Self-reported questionnaire measured acceptability of all elements of intervention delivery

SECONDARY OUTCOMES:
Objectively-measured incidental physical activity | Change from baseline to 13 weeks
  Minutes spent in activity per day measured using the activPAL device.
Participant questionnaire reported motivation: 15 item Likert scale | Change from baseline to 13 weeks
  15 item scale adapted from Markland, D. & Tobin, V. (2004). Journal of Sport and Exercise Psychology, 26, 191-196 (BREQ-2 for PA)
Participant questionnaire measured work-related productivity: Likert scale | Change from baseline to 13 weeks
  Likert scale of productivity adapted from Kessler et al's World Health Organisation Health and Work Performance Questionnaire (HPQ)
Participant self-reported monthly cycling activity: number of rides and duration | Change from baseline to 13 weeks
  Questionnaire measured of cycling activity adapted from Craig CL, Marshall AL, Sjostrom M, Bauman A, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P: International Physical Activity Questionnaire: 12-country reliability and validity. Medicine and Science in Sports and Exercise 2003, 35:1381-1395.
  Craig CL, Marshall AL, Sjostrom M, Bauman A, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P: International Physical Activity Questionnaire: 12-country reliability and validity. Medicine and Science in Sports and Exercise 2003, 35:1381-1395.
  Adapted DINE questionnaire: Roe L, Strong C, Whiteside C, Neil A, Mant D. Dietary intervention in primary care: validity of the DINE method for diet assessment. Fam Pract 1994; 11: 375-81.
Participant self-reported dietry intake: DINE questionnaire | Change from baseline to 13 weeks
  Adapted DINE questionnaire: Roe L, Strong C, Whiteside C, Neil A, Mant D. Dietary intervention in primary care: validity of the DINE method for diet assessment. Fam Pract 1994; 11: 375-81.
Participant self-reported number of days of work-related absenteeism/presenteeism | Change from baseline to 13 weeks
  Self reported days per month of absenteeism/presenteeism adapted from Kessler et al's World Health Organisation Health and Work Performance Questionnaire (HPQ)
Participant self reported job satisfaction: Likert scale | Change from baseline to 13 weeks
  Questionnaire measured job satisfaction adapted from Kessler et al's World Health Organisation Health and Work Performance Questionnaire (HPQ)
Participant self-reported work-related stress: Likert scale | Change from baseline to 13 weeks
  Questionnaire measured work-related stress adapted from Kessler et al's World Health Organisation Health and Work Performance Questionnaire (HPQ)
Participant self-reported autonomy: Likert scale | Change from baseline to 13 weeks
  Questionnaire measured autonomy adapted from Bartholomew, K. J., Ntoumanis, N., Ryan, R. M., & Thøgersen-Ntoumani, C. (2011). Journal of Sport & Exercise Psychology, 33, 75e102.
Participant self-reported competence: 6 item Likert scale | Change from baseline to 13 weeks
  Questionnaire measured competence adapted from Roberts, G.C., Treasure D. C., & Balague, G. (1998). Achievement goals in sport: The development and validation of the Perception of Success Questionnaire. Journal of Sport Sciences. 19, 337-347.
Participant self-reported relatedness: 6 item Likert scale | Change from baseline to 13 weeks
  Questionnaire measured relatedness adapted from Van den Broeck et al (2010). J Occup Organiz Psych 83:981-1002
Participant self-reported perceptions of cycling safety: 5 item Likert scale | Change from baseline to 13 weeks
  Questionnaire measured scale of perceptions of cycling safety
Participant self-reported wellbeing: 14 item Warwick-Edinburgh Mental Wellbeing Scales - WEMWBS | Change from baseline to 13 weeks
  Questionnaire measured participant wellbeing.
Participant self-reported self esteem: 10 item Rosenberg scale of self esteem | Change from baseline to 13 weeks
  Self-esteem questionnaire
Participant self-reported vitality: 4 item Bostic scale | Change from baseline to 13 weeks
  4-item scale of vitality (Bostic, T. J., McGartland-Rubio, D., & Hood, M. (2000). A validation of the subjective vitality scale using structural equation modeling)
Participant self-reported general physical health: EQ-5D-5L | Change from baseline to 13 weeks
  Questionnaire measure of health-related quality of life
Body mass | Change from baseline to 13 weeks
  Body mass in kilograms
Body Mass Index (BMI) | Change from baseline to 13 weeks
  Weight and height will be combined to report BMI in kg/m^2
Waist circumference | Change from baseline to 13 weeks
  Waist circumference in centimeters

OTHER OUTCOMES:
Blood pressure | Change from baseline to 13 weeks
Homestasis Model Estimated Insulin Resistance (HOMA-IR) | Change from baseline to 13 weeks
  Calculated from fasting insulin and glucose concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Jason MR Gill, PhD, Principal Investigator — University of Glasgow; Cindy M Gray, PhD, Principal Investigator — University of Glasgow
Locations (1):
- University of Glasgow, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No
These data will only be handled by UoG researchers

REFERENCES:
- [Background] Kelly P, Kahlmeier S, Gotschi T, Orsini N, Richards J, Roberts N, Scarborough P, Foster C. Systematic review and meta-analysis of reduction in all-cause mortality from walking and cycling and shape of dose response relationship. Int J Behav Nutr Phys Act. 2014 Oct 24;11:132. doi: 10.1186/s12966-014-0132-x. PMID 25344355
- [Background] Sahlqvist S, Goodman A, Simmons RK, Khaw KT, Cavill N, Foster C, Luben R, Wareham NJ, Ogilvie D. The association of cycling with all-cause, cardiovascular and cancer mortality: findings from the population-based EPIC-Norfolk cohort. BMJ Open. 2013 Nov 14;3(11):e003797. doi: 10.1136/bmjopen-2013-003797. PMID 24231462
- [Background] Schnohr P, Marott JL, Jensen JS, Jensen GB. Intensity versus duration of cycling, impact on all-cause and coronary heart disease mortality: the Copenhagen City Heart Study. Eur J Prev Cardiol. 2012 Feb;19(1):73-80. doi: 10.1177/1741826710393196. Epub 2011 Feb 21. PMID 21450618
- [Background] Andersen LB, Schnohr P, Schroll M, Hein HO. All-cause mortality associated with physical activity during leisure time, work, sports, and cycling to work. Arch Intern Med. 2000 Jun 12;160(11):1621-8. doi: 10.1001/archinte.160.11.1621. PMID 10847255
- [Background] Oja P, Kelly P, Pedisic Z, Titze S, Bauman A, Foster C, Hamer M, Hillsdon M, Stamatakis E. Associations of specific types of sports and exercise with all-cause and cardiovascular-disease mortality: a cohort study of 80 306 British adults. Br J Sports Med. 2017 May;51(10):812-817. doi: 10.1136/bjsports-2016-096822. Epub 2016 Nov 28. PMID 27895075
- [Background] Celis-Morales CA, Lyall DM, Welsh P, Anderson J, Steell L, Guo Y, Maldonado R, Mackay DF, Pell JP, Sattar N, Gill JMR. Association between active commuting and incident cardiovascular disease, cancer, and mortality: prospective cohort study. BMJ. 2017 Apr 19;357:j1456. doi: 10.1136/bmj.j1456. PMID 28424154
- [Background] Blond K, Jensen MK, Rasmussen MG, Overvad K, Tjonneland A, Ostergaard L, Grontved A. Prospective Study of Bicycling and Risk of Coronary Heart Disease in Danish Men and Women. Circulation. 2016 Nov 1;134(18):1409-1411. doi: 10.1161/CIRCULATIONAHA.116.024651. No abstract available. PMID 27799259
- [Background] Kubesch NJ, Therming Jorgensen J, Hoffmann B, Loft S, Nieuwenhuijsen MJ, Raaschou-Nielsen O, Pedersen M, Hertel O, Overvad K, Tjonneland A, Prescot E, Andersen ZJ. Effects of Leisure-Time and Transport-Related Physical Activities on the Risk of Incident and Recurrent Myocardial Infarction and Interaction With Traffic-Related Air Pollution: A Cohort Study. J Am Heart Assoc. 2018 Jul 18;7(15):e009554. doi: 10.1161/JAHA.118.009554. PMID 30021805
- [Background] Hoevenaar-Blom MP, Wendel-Vos GC, Spijkerman AM, Kromhout D, Verschuren WM. Cycling and sports, but not walking, are associated with 10-year cardiovascular disease incidence: the MORGEN Study. Eur J Cardiovasc Prev Rehabil. 2011 Feb;18(1):41-7. doi: 10.1097/HJR.0b013e32833bfc87. PMID 20543701
- [Background] Tanasescu M, Leitzmann MF, Rimm EB, Willett WC, Stampfer MJ, Hu FB. Exercise type and intensity in relation to coronary heart disease in men. JAMA. 2002 Oct 23-30;288(16):1994-2000. doi: 10.1001/jama.288.16.1994. PMID 12387651
- [Background] Millett C, Agrawal S, Sullivan R, Vaz M, Kurpad A, Bharathi AV, Prabhakaran D, Reddy KS, Kinra S, Smith GD, Ebrahim S; Indian Migration Study group. Associations between active travel to work and overweight, hypertension, and diabetes in India: a cross-sectional study. PLoS Med. 2013;10(6):e1001459. doi: 10.1371/journal.pmed.1001459. Epub 2013 Jun 11. PMID 23776412
- [Background] Laverty AA, Mindell JS, Webb EA, Millett C. Active travel to work and cardiovascular risk factors in the United Kingdom. Am J Prev Med. 2013 Sep;45(3):282-8. doi: 10.1016/j.amepre.2013.04.012. PMID 23953354
- [Background] Rasmussen MG, Grontved A, Blond K, Overvad K, Tjonneland A, Jensen MK, Ostergaard L. Associations between Recreational and Commuter Cycling, Changes in Cycling, and Type 2 Diabetes Risk: A Cohort Study of Danish Men and Women. PLoS Med. 2016 Jul 12;13(7):e1002076. doi: 10.1371/journal.pmed.1002076. eCollection 2016 Jul. PMID 27403867
- [Background] Mytton OT, Ogilvie D, Griffin S, Brage S, Wareham N, Panter J. Associations of active commuting with body fat and visceral adipose tissue: A cross-sectional population based study in the UK. Prev Med. 2018 Jan;106:86-93. doi: 10.1016/j.ypmed.2017.10.017. Epub 2017 Oct 10. PMID 29030265
- [Background] Hollingworth M, Harper A, Hamer M. Dose-response associations between cycling activity and risk of hypertension in regular cyclists: The UK Cycling for Health Study. J Hum Hypertens. 2015 Apr;29(4):219-23. doi: 10.1038/jhh.2014.89. Epub 2014 Oct 2. PMID 25273856
- [Background] Rasmussen MG, Overvad K, Tjonneland A, Jensen MK, Ostergaard L, Grontved A. Changes in Cycling and Incidence of Overweight and Obesity among Danish Men and Women. Med Sci Sports Exerc. 2018 Jul;50(7):1413-1421. doi: 10.1249/MSS.0000000000001577. PMID 29443821
- [Background] Oja P, Titze S, Bauman A, de Geus B, Krenn P, Reger-Nash B, Kohlberger T. Health benefits of cycling: a systematic review. Scand J Med Sci Sports. 2011 Aug;21(4):496-509. doi: 10.1111/j.1600-0838.2011.01299.x. Epub 2011 Apr 18. PMID 21496106
- [Background] de Geus B, Van Hoof E, Aerts I, Meeusen R. Cycling to work: influence on indexes of health in untrained men and women in Flanders. Coronary heart disease and quality of life. Scand J Med Sci Sports. 2008 Aug;18(4):498-510. doi: 10.1111/j.1600-0838.2007.00729.x. Epub 2007 Dec 7. PMID 18067515
- [Background] Moller NC, Ostergaard L, Gade JR, Nielsen JL, Andersen LB. The effect on cardiorespiratory fitness after an 8-week period of commuter cycling--a randomized controlled study in adults. Prev Med. 2011 Sep;53(3):172-7. doi: 10.1016/j.ypmed.2011.06.007. Epub 2011 Jun 25. PMID 21708185
- [Background] Crane M, Rissel C, Standen C, Greaves S. Associations between the frequency of cycling and domains of quality of life. Health Promot J Austr. 2014 Dec;25(3):182-5. doi: 10.1071/HE14053. PMID 25481703
- [Background] Mytton OT, Panter J, Ogilvie D. Longitudinal associations of active commuting with wellbeing and sickness absence. Prev Med. 2016 Mar;84:19-26. doi: 10.1016/j.ypmed.2015.12.010. Epub 2015 Dec 29. PMID 26740344
- [Background] Rojas-Rueda D, de Nazelle A, Tainio M, Nieuwenhuijsen MJ. The health risks and benefits of cycling in urban environments compared with car use: health impact assessment study. BMJ. 2011 Aug 4;343:d4521. doi: 10.1136/bmj.d4521. PMID 21816732
- [Background] Stewart G, Anokye NK, Pokhrel S. What interventions increase commuter cycling? A systematic review. BMJ Open. 2015 Aug 14;5(8):e007945. doi: 10.1136/bmjopen-2015-007945. PMID 26275902
- [Background] Bird EL, Baker G, Mutrie N, Ogilvie D, Sahlqvist S, Powell J. Behavior change techniques used to promote walking and cycling: a systematic review. Health Psychol. 2013 Aug;32(8):829-38. doi: 10.1037/a0032078. Epub 2013 Mar 11. PMID 23477577